Protocol cover page NCT03274076

EVALUATION OF TOFACITINIB IN EARLY DIFFUSE CUTANEOUS SYSTEMIC SCLEROSIS: A PHASE I/II TWO-CENTER SAFETY AND TOLERABILITY STUDY

Date: March 2019

# Evaluation of Tofacitinib in Early Diffuse Cutaneous Systemic Sclerosis: A Phase I/II Two-Center Safety and Tolerability Study Final Statistical Analysis Plan

Statistical Author: Jeff Moore, MS

Principal Investigator: Dinesh Khanna, MD

# Contents

| 1.1. Primary Endpoint | 5 |
|---|---|
| <ol> <li>Secondary Analysis of the Primary Endpoint.</li> <li>Secondary Endpoints</li></ol> | 5 |
| 1.2.1. Secondary Endpoint. Analyses of the Primary Endpoint Over Time 1.2.2. Secondary Endpoint. Analyses of the Adverse Events at the Grade 2 | 5 |
| <ul><li>1.2.1. Secondary Endpoint. Analyses of the Primary Endpoint Over Time</li><li>1.2.2. Secondary Endpoint. Analyses of the Adverse Events at the Grade 2</li></ul> | 5 |
| 1.2.2. Secondary Endpoint. Analyses of the Adverse Events at the Grade 2 | 5 |
| | 5 |
| 1 2 2 Secondary Endnoint % of Subjects with Adverse Events of Special In | Threshold6 |
| 1.2.3. Secondary Enapoint. % of Subjects with Adverse Events of Special III | terest (AESI)6 |
| 1.2.4. Secondary Endpoint. Change from Baseline in the Modified Rodnan | Skin Score (mRSS)6 |
| 1.2.5. Secondary Endpoint. Provisional American College of Rheumatology | Combined Response Index in Systemic Sclerosis 6 |
| 1.2.6. Secondary Endpoint. % of Responders as Defined by the mRSS | 6 |
| 1.2.7. Secondary Endpoint. Change from Baseline in the mRSS sub-scores. | 6 |
| 1.2.8. Secondary Endpoint. Change from Baseline in Physician Global Heal | th Assessment7 |
| 1.2.9. Secondary Endpoint. Change from Baseline in Patient Global Health | Assessment7 |
| 1.2.10. Secondary Endpoint. Change from Baseline in Health Related Qua Outcomes Measurement Information System (PROMIS-29) | |
| 1.2.11. Secondary Endpoint. Change from Baseline in the Scleroderma He (SHAQ-DI) | |
| 1.2.12. Secondary Endpoint. Change from Baseline in the UCLA SCTC Gast | trointestinal Symptoms Total Score (GIT)7 |
| <ul><li>1.2.13. Secondary Endpoint. Change from Baseline in the PRO for Sclerod</li><li>Score. 7</li></ul> | erma-related Skin Symptoms (PRO-SRSS) Total |

| | 1.2.14. | Secondary Endpoint. Change from Screening in Pulmonary Function Tests (PFT) | 8 |
|---|---|---|---|
| | 1.2.15.<br>Range). | Secondary Endpoint. Change from Screening to Week 24 in Left Ventricular Ejection Fraction (Maximum of 8 | |
| | 1.2.16. | Secondary Endpoint. Change from Screening to Week 24 in Tricuspid Regurgitation Jet | 8 |
| | 1.3. Expl | oratory Endpoints | 8 |
| | 1.4. Add | itional Measures | 8 |
| 2. | Analysi | is Strategy | 8 |
| | | ly Populations | |
| | 2.2. Ana | lyses of Primary Endpoint | 9 |
| | 2.2.1. | Primary Analysis of the Primary Endpoint | 9 |
| | 2.2.2. | Secondary Analysis of the Primary Endpoint | 10 |
| | 2.3. Ana | lyses of Secondary Endpoints | 10 |
| | 2.3.1. | Analyses of the primary endpoint over time | 10 |
| | 2.3.2. | Secondary analyses of the primary endpoint over time | 11 |
| | 2.3.3. | Secondary analyses for proportion of subjects | 11 |
| | 2.3.4. | Secondary analyses for continuous endpoints | 12 |
| | 2.4. Ana | lyses of Exploratory Endpoints | 13 |
| 3. | Table, | Listing and Figure Shells | 13 |
| | 3.1.1. | Subject Characteristics and Study Conduct | 13 |
| | 3.1.2. | Safety Analyses | 31 |
| | 3.1.3. | Efficacy Analyses | 117 |

#### 1. Endpoints and Other Outcomes

This section describes the primary and secondary efficacy outcomes, as well as safety and other outcomes.

## 1.1. Primary Endpoint

**Objective**: To demonstrate acceptable safety and tolerability of tofacitinib in early dcSSc.

The primary endpoint is the proportion of participants who experience Grade 3 or higher (more severe) adverse events that occur at or before Week 24 (double-blind phase).

#### 1.1.1. Primary Analysis of the Primary Endpoint.

The proportion of subjects in the safety population (see Section 2.1) with at least one Grade 3 or higher adverse event that begins at or before Week 24, the double-blind phase of the trial, will be calculated and compared for each of the study treatment arms.

#### 1.1.2. Secondary Analysis of the Primary Endpoint.

To assess the robustness of the results for the primary analysis, an analysis of the total number of Grade 3 (severe) or higher adverse events that begin at or before Week 24 will also be compared for each of the study treatment arms.

# 1.2. Secondary Endpoints

# **1.2.1.** Secondary Endpoint. Analyses of the Primary Endpoint Over Time.

The analyses of the primary endpoint described in sections 1.1.1 and 1.1.2 will be repeated at Weeks 12 to assess the time course of the safety profile as defined by the occurrence of Grade 3 or higher adverse events.

#### 1.2.2. Secondary Endpoint. Analyses of the Adverse Events at the Grade 2 Threshold.

The analyses described in sections 1.1.1, 1.1.2 and 1.2.1 will be repeated for adverse events beginning at or before the time point of interest that are assessed as at least Grade 2 (moderate) severity.

#### 1.2.3. Secondary Endpoint. % of Subjects with Adverse Events of Special Interest (AESI).

The proportion of subjects in the safety population experiencing an AESI will be compared between the two study treatment arms. Comparisons will be made for at least one AESI of any type, as well as for each of the events that are considered to be of special interest individually. Separate analyses will be performed for AESIs that occur at or before Weeks 12 and 24. AESIs are defined to be any one of herpes zoster, malignancy, serious infection, lymphocytes <500cells mm³, ANC <500cells mm³, AST > 3xULN, ALT > 3xULN, Hy's Law criteria met, Hemoglobin drop > 2mg/dL, increase in HDL/LDL ratio > 50%, or an increase in serum creatinine > 50%.

#### 1.2.4. Secondary Endpoint. Change from Baseline in the Modified Rodnan Skin Score (mRSS).

Change from baseline in the mRSS total score will be compared between the two treatment arms to assess skin thickness relative to the initiation of study treatment at the various time points. The analysis will be performed separately at Weeks 12 and 24 on subjects in the modified intent-to-treat (mITT) population (see section 2.1).

1.2.5. Secondary Endpoint. Provisional American College of Rheumatology Combined Response Index in Systemic Sclerosis CRISS will be compared between the two treatment arms separately at Weeks 12 and 24 on subjects in the modified intent-to-treat (mITT) population (see section 2.1).

#### 1.2.6. Secondary Endpoint. % of Responders as Defined by the mRSS.

Subjects in the mITT population will be assessed for reaching clinical thresholds of decreased skin thickness over time as defined by a percentage reduction in the mRSS from baseline. Time points assessed will be Weeks 12 and 24, and analyzed separately. Within each of these time points, separate analyses will be performed for decreases (responder definition) of at least 20, 40, and 60% relative to the baseline mRSS total score.

#### 1.2.7. Secondary Endpoint. Change from Baseline in the mRSS sub-scores.

Change from baseline in the mRSS representative score and maximum score will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately.

#### 1.2.8. Secondary Endpoint. Change from Baseline in Physician Global Health Assessment.

Change from baseline in the physician's global health assessment will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately, to determine overall progression of disease severity as determined by the subject's physician.

#### 1.2.9. Secondary Endpoint. Change from Baseline in Patient Global Health Assessment.

Change from baseline in the patient's global health assessment will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately, to determine overall progression of disease severity as determined by the subject.

# 1.2.10. Secondary Endpoint. Change from Baseline in Health Related Quality of Life (HRQoL) using the Patient-Reported Outcomes Measurement Information System (PROMIS-29).

Change from baseline in the HRQoL total score will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately to determine perceived overall changes in quality of life since the initiation of study treatment as determined by the subject.

# 1.2.11. Secondary Endpoint. Change from Baseline in the Scleroderma Health Assessment Questionnaire-Disability Index (SHAQ-DI).

Change from baseline in the SHAQ-DI total score will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately to determine perceived overall changes in the subject's functional ability since the initiation of study treatment as determined by the subject.

#### 1.2.12. Secondary Endpoint. Change from Baseline in the UCLA SCTC Gastrointestinal Symptoms Total Score (GIT).

Change from baseline in the UCLA SCTC GIT will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately to determine changes in the subject's gastrointestinal symptoms since the initiation of study treatment.

### 1.2.13. Secondary Endpoint. Change from Baseline in the PRO for Scleroderma-related Skin Symptoms (PRO-SRSS) Total Score.

Change from baseline in the PRO-SRSS will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately to determine changes in the subject's overall skin symptoms since the initiation of study treatment.

#### 1.2.14. Secondary Endpoint. Change from Screening in Pulmonary Function Tests (PFT).

Change from screening PFTs will be compared between the two study treatment arms for the mITT population of subjects at Weeks 12 and 24 separately for each of percent predicted FVC, FEV and DLCO.

#### 1.2.15. Secondary Endpoint. Change from Screening to Week 24 in Left Ventricular Ejection Fraction (Maximum of Range).

Change from screening ejection fraction will be compared between the two study treatment arms for the mITT population of subjects at Week 24.

#### 1.2.16. Secondary Endpoint. Change from Screening to Week 24 in Tricuspid Regurgitation Jet.

Change from screening tricuspid regurgitation jet will be compared between the two study treatment arms for the mITT population of subjects at Week 24.

#### 1.3. Exploratory Endpoints

Analyses of each of the secondary endpoints will be provided at weeks 36 and 48, provided the item was collected.

#### 1.4. Additional Measures

Additionally, the following measures will be provided descriptively (no inferential analyses) by study treatment arm for the safety population:

- Clinical laboratory values over time.
- Vital signs over time.
- Physical examination findings.
- Concomitant medication.

# 2. Analysis Strategy

No formal interim analyses of the primary endpoint were conducted, therefore the nominal  $\alpha$  level to be used at the final analysis is 0.10 for the primary endpoint. All other secondary outcomes will also be tested at the 10% level, with no adjustment for multiplicity. Given the limited statistical power for a study consisting of 15 subjects, models will not include covariates.

# 2.1. Study Populations

Two study populations will be defined for these analyses:

- **Modified Intent to Treat (mITT):** The mITT analysis set consists of all subjects randomized, receiving at least one dose of treatment, and having at least one post-baseline efficacy assessment for the given parameter. No imputation techniques will be utilized for missing observations.
- Safety: The safety population consists of all subjects who were randomized and received at least one dose of the study drug.

#### 2.2. Analyses of Primary Endpoint

The primary analysis is a comparison of the percentage of subjects with Grade 3 adverse events that begin within the first 24 Weeks following initiation of study treatment between tofacitinib and placebo. The analysis will be performed on the safety population. The test will be performed using Fisher's Exact Test, given that the largest possible number of patients affected are 10 and 5, respectively, for tofacitinib and placebo. The number and percentage of patients with at least one Grade 3 adverse event will be provided along with Clopper Pearson Exact confidence intervals for proportions at the 90% threshold.

#### 2.2.1. Primary Analysis of the Primary Endpoint.

Proportion of patients with at least one Grade 3 adverse event within the first 24 Weeks

| Analysis Set | Safety Population |
|---|---|
| Methods | Fisher's Exact Test |
| | Clopper Pearson Exact Confidence Intervals |
| Results | <ul> <li>Number and percentage of subjects with at least one Grade 3 adverse event in the first 24 weeks</li> <li>90% confidence interval for proportions</li> <li>P-value from Fisher's Exact Test</li> </ul> |

#### 2.2.2. Secondary Analysis of the Primary Endpoint.

A sensitivity analysis will be performed to assess how the total number of Grade 3 or higher adverse events, rather than just the proportion of patients experiencing the events, affect the conclusions of the analysis of the primary endpoint. The analysis will employ Poisson Regression methodology, offset for time in the study (the lesser of 24 weeks, or withdrawal from the trial).

| Analysis Set | Safety Population |
|---|---|
| Methods | Poisson Regression offset for time in the study (the lesser of 24 weeks or |
| | withdrawal from the trial) |
| Dependent | Number of grade 3 or higher adverse events experienced within the first |
| Variable | 24 weeks on a per patient basis. |
| Covariate | Treatment |
| Results • Total number of Grade 3 adverse event in the first 24 week | |
| | <ul> <li>Relative risk of tofacitinib to placebo.</li> </ul> |
| | <ul> <li>90% confidence interval for relative risk</li> </ul> |
| | P-value for treatment effect |

# 2.3. Analyses of Secondary Endpoints

#### 2.3.1. Analyses of the primary endpoint over time.

The secondary analyses is a comparison of the percentage of subjects with Grade 3 adverse events that begin within the first 12, 36, and 48 Weeks, respectively, following initiation of study treatment between tofacitinib and placebo. Each of the time points is a standalone analysis, utilizing the methodology described for the primary analysis of the primary endpoint in section 2.2.1

| Analysis Set | Safety Population |
|-----------------------------|--------------------------------------------|
| Time Points | 2.3.1a: Week 12, |
| | 2.3.1b: Week 36, |
| | 2.3.1c: Week 46 |
| Methods Fisher's Exact Test | |
| | Clopper Pearson Exact Confidence Intervals |

| Results | • | Number and percentage of subjects with at least one Grade 3 |
|---|---|---|
| adverse event up to and including the time point of ir | | adverse event up to and including the time point of interest |
| | • | 90% confidence interval for proportions |
| | • | P-value from Fisher's Exact Test |

#### 2.3.2. Secondary analyses of the primary endpoint over time.

Secondary analyses will be performed over time (Weeks 12, 36 and 48) using the same methodology described in section 2.2.2 to explore treatment differences in the total number of Grade 3 or higher adverse events over time. The offset for time in study will be the lesser of the withdrawal date from the trial or the time point of interest.

| Analysis Set | Safety Population |
|---|---|
| Methods | Poisson Regression offset for time in the study (the lesser of the time |
| | point of interest or withdrawal from the trial) |
| Time Points | 2.3.2a: Week 12, |
| | 2.3.2b: Week 36, |
| | 2.3.2c: Week 46 |
| Dependent | Number of grade 3 or higher adverse events experienced within the time |
| Variable | point of interest on a per patient basis. |
| Covariate | Treatment |
| Results | Total number of Grade 3 adverse event within the time point of |
| interest. | |
| | Relative risk of tofacitinib to placebo. |
| | 90% confidence interval for relative risk |
| | P-value for treatment effect |

#### 2.3.3. Secondary analyses for proportion of subjects.

The proportion of subjects in the specified populations above will be compared between the two study treatment arms at the specified time points utilizing Fisher's Exact Test and Clopper Pearson confidence intervals to describe treatment differences.

| Analysis Set | See Above |
|--------------|-----------|
| Time Points | See Above |

| Parameters | Adverse events of special interest |
|---|---|
| | mRSS responders |
| Methods | Fisher's Exact Test |
| | Clopper Pearson Exact Confidence Intervals |
| Results • Number and percentage of subjects with at the parameter of subjects with a subject subject subject subject subjects. | |
| | interest. |
| | <ul> <li>90% confidence interval for proportions</li> </ul> |
| | P-value from Fisher's Exact Test |

## 2.3.4. Secondary analyses for continuous endpoints.

Continuous parameters will be analyzed utilizing a two-sample t-test to explore treatment differences at the time points described above. There will be no further adjustments. Descriptive statistics (e.g. mean, standard deviation, median, min, and max) will be provided by treatment to further describe the distributions. If there are specific concerns about outliers, suggesting a skewed distribution, a Wilcoxon Rank Sum test will be additionally provided as a sensitivity analysis.

| Analysis Set | See Above |
|---|---|
| Time Points | See Above |
| Parameters | <ul> <li>Change from baseline in mRSS total score.</li> </ul> |
| | <ul> <li>CRISS scores at Weeks 12 and 24.</li> </ul> |
| | <ul> <li>Change from baseline in physician's global health assessment.</li> </ul> |
| | <ul> <li>Change from Baseline in Patient Global Health Assessment.</li> </ul> |
| | <ul> <li>Change from Baseline in Health Related Quality of Life (HRQoL).</li> </ul> |
| | Change from Baseline in the Scleroderma Health Assessment |
| | Questionnaire-Disability Index (SHAQ-DI). |
| | <ul> <li>Change from Baseline in the UCLA SCTC Gastrointestinal</li> </ul> |
| | Symptoms Total Score (GIT). |
| | <ul> <li>Change from Baseline in the PRO for Scleroderma-related Skin</li> </ul> |
| | Symptoms (PRO-SRSS) Total Score. |
| | <ul> <li>Change from Screening in Pulmonary Function Tests (PFT) – FVC,</li> </ul> |
| | FEV and DLCO. |
| | <ul> <li>Secondary Endpoint. Change from Screening to Week 24 in Left</li> </ul> |
| | Ventricular Ejection Fraction (Maximum of Range). |

| | <ul> <li>Change from screening ejection fraction will be compared between the two study treatment arms for the mITT population of subjects at Week 24.</li> <li>Secondary Endpoint. Change from Screening to Week 24 in Tricuspid Regurgitation Jet.</li> <li>Change from screening tricuspid regurgitation jet will be compared between the two study treatment arms for the mITT population of subjects at Week 24.</li> </ul> |
|---|---|
| Methods | Two sample t-test |
| Results | Mean |
| | Standard deviation |
| | Median |
| | Min, Max |
| | P-value from t-test |

# 2.4. Analyses of Exploratory Endpoints

Each of the items above will be analyzed for weeks 36 and 48 using the methodology described for the given time, provided the item was collected at these time points.

# 3. Table, Listing and Figure Shells

Note: Weeks 36 and 48 are exploratory, and will be provided in separate, supplemental tables following the reporting of primary and secondary endpoints.

# 3.1.1. Subject Characteristics and Study Conduct

**Table 1: TOFA Subject Disposition. All Subjects** 

| Status | Tofacitinib<br>N (%) | Placebo<br>N (%) |
|---|---|---|
| ITT Population [1] | | |
| Safety Population [2] | | |
| Open Label Population [3] | | |
| Completed Study Treatment | | |
| Discontinued Study Early | | |
| Reason for Discontinuation | | |
| Subject was determined to be ineligible | | |
| Subject withdrew consent | | |
| Investigator withdrew subject | | |
| Study terminated by Sponsor | | |
| Death | | |
| Lost to follow-up | | |
| Other | | |
| Permanently Discontinued Study Treatment | | |
| Reason for Discontinuation of Study Treatment | | |
| Adverse Event | | |

Note: Percentages are based on the number of subjects in the Safety Population.

- [1] The ITT population includes all patients randomized to TOFA.
- [2] The Safety Population includes all randomized subjects who received at least one dose of study medication.
- [3] The Open Label Population includes all patients in the Safety Population that have completed 24 weeks (168 Days) of Double-Blind study treatment and not withdrawn from the study.

Data cutoff date: DDMMYY

**Listing 1: TOFA Early Termination. ITT Subjects.** 

| Subject<br>ID | Treatment | Reason for<br>Discontinuation | Time on Treatment (Days) | Time in Study (Days) |
|---|---|---|---|---|

Conditional Note: No patients have discontinued as of the data cutoff date.

**Table 2: TOFA Demographic Characteristics. ITT Population** 

| Variable<br>Statistic or Category | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----------------------------------|---------------------|----------------|
| Age (Years) | | |
| N | | |
| Mean | | |
| SD | | |

| | Tofacitinib | Placebo |
|-----------------------------------|-------------|---------|
| Variable<br>Statistic or Category | N=10 | N=5 |
| Median | 11 20 | 11 0 |
| Min, Max | | |
| Age, n (%) | | |
| 18 to 35 years | | |
| >35 to 55 years | | |
| >55 to 70 years | | |
| Gender, n (%) | | |
| Male | | |
| Female | | |
| Of Childbearing Age | | |
| Not of Childbearing Age | | |
| Hysterectomy | | |
| Tubal Ligation | | |
| Post Menopausal | | |
| Other Reason | | |
| Ethnicity, n (%) | | |
| Hispanic or Latino | | |
| Not Hispanic or Latino | | |
| Race, n (%) [1] | | |
| American Indian or Alaska Native | | |
| Asian | | |

| Variable<br>Statistic or Category | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|
| Black or African-American | | |
| Native Hawaiian or Other Pacific Islander | | |
| White | | |
| Not Reported | | |
| Smoking History, n (%) [1] | | |
| Never | | |
| Past History | | |
| Current Smoker | | |
| No Response | | |

Note: Percentages are 100\*n/N

[1] Subjects reporting more than one race are counted in each of the race categories reported.

**Table 3: TOFA Baseline Characteristics. ITT Population** 

| Variable<br>Statistic or Category | Tofacitinib<br>N = 10 | Placebo<br>N = 5 |
|-----------------------------------|-----------------------|------------------|
| mRss at Baseline | | |
| N | | |

| Variable<br>Statistic or Category | Tofacitinib<br>N = 10 | Placebo<br>N = 5 |
|---|---|---|
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Disease Duration Since 1st Non-Raynaud's Sign or Symptom (Years) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Disease Duration Since Raynaud's Phenomenon (Years) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Interstitial lung disease on HRCT of chest, N (%) | | |
| FVC% - at Screening | | |
| N | | |
| Mean | | |

| Variable<br>Statistic or Category | Tofacitinib<br>N = 10 | Placebo<br>N = 5 |
|---|---|---|
| SD | | |
| Median | | |
| Min, Max | | |
| DLCO% - at Screening | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| HAQ-DI [theoretical range, 0-3] | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| SHAQ: Pain From Illness in Past Week (theoretical range, 0-150) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |

| Variable<br>Statistic or Category | Tofacitinib<br>N = 10 | Placebo<br>N = 5 |
|---|---|---|
| Min, Max | | |
| SHAQ: Intestinal Problems Interfere with Daily Activities in Past Week [theoretical range, 0-150] | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| SHAQ: Breathing Problems Interfere with Daily Activities in Past Week [theoretical range, 0-150] | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| SHAQ: Raynaud's Interfere with Daily Activities in Past Week [theoretical range, 0-150] | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |

| Variable | Tofacitinib | Placebo |
|---|---|---|
| Statistic or Category | N = 10 | N = 5 |
| Min, Max | | |
| SHAQ: Finger Ulcers Interfere with Daily Activities in Past Week [theoretical range, 0-150] | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Hemoglobin (g/dL) - at Screening | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| WBC (K/uL) - at screening | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Large Joint Contracture N (%) | | |

| Variable<br>Statistic or Category | Tofacitinib<br>N = 10 | Placebo<br>N = 5 |
|---|---|---|
| Small Joint Contracture N (%) | | |
| Tendon Friction Rub (Range 0 to 12) ** | | |
| # (%) with 0 positive results | | |
| # (%) with 1 positive result | | |
| # (%) with 2 positive results | | |
| # (%) with ANY positive results | | |

**Table 4: TOFA Baseline ECHO. ITT Population** 

| Variable<br>Statistic or Category | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|
| Left Ejection Fraction (Maximum of Range) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |

<sup>\*\*</sup> Areas of examination include right and left shoulder, elbow, wrist, MCP, knee, and ankle.

| Variable<br>Statistic or Category | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|
| Min, Max | | |
| EV Enlargement: N (%) | | |
| Right Ventricular Diameter For Patients with Enlargement (mm) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| RVSP: N (%) | | |
| RVSP Value (mmHg) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Pericardial Effusion Moderate to Large: N (%) | | |

**Table 5: TOFA Study Drug Compliance. ITT Population** 

| Variable<br>Statistic or Category | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|
| Study Drug Exposure (Days) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Study Drug Compliance % (Actual Tablets Used/Expected Tablets Used) | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min, Max | | |
| Study Drug Compliance % Thresholds for Dosed Subjects | | |
| Number of Subjects Dosed | | |
| < 75% | | |
| 75-85% | | |
| 85-95% | | |
| 95-99% | | |

| Variable<br>Statistic or Category | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----------------------------------|---------------------|----------------|
| 100% | | |
| 101-105% | | |
| At least 95% Compliant | | |

Table 6: TOFA Summary of Immunosuppressive Therapy. Safety Population

| Variable | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|
| # of Subjects | | |
| # of Subjects with Immunosuppressive<br>Therapy | | |
| % of Subjects with Immunosuppressive<br>Therapy | | |

**Listing 2: Immunosuppressive Therapy. Safety Population** 

| Treatment | Subject<br>ID | Medication | Start Date | Stop<br>Date | Medicatio<br>n Ongoing |
|---|---|---|---|---|---|

**Table 7: TOFA Concomitant Medication Usage. Safety Population [1]** 

| <b>Concomitant Medication</b> | Tofacitinib N=10 n(%) | Placebo N=5<br>n(%) |
|-------------------------------|-----------------------|---------------------|
| Abreva | | |
| Acyclovir | | |
| Adderall XR | | |
| Aleve | | |
| Amlodipine(Norvasc) | | |
| Asprin | | |
| Atorvastatin(Lipitor) | | |
| Augmentin | | |
| Bydureon | | |
| Calcium with Vitamin D | | |
| Carafate | | |
| Celebrex | | |
| Ciprofloxacin(Cipro) | | |
| Clindamycin(Cleocin) | | |
| Clonazepam(Klonopin) | | |
| CoQ10 | | |
| Collagenase | | |
| Compezine | | |
| Cymbalta | | |

| Concomitant Medication | Tofacitinib N=10 n(%) | Placebo N=5<br>n(%) |
|---|---|---|
| Diazepam(Valium) | | |
| Diltiazem | | |
| Duloxetine(Cymbalta) | | |
| Esomeprazole magnesium(Nexium) | | |
| Ferrous Sulfate | | |
| Flexeril | | |
| Flonase | | |
| Folic Acid | | |
| Furosemide(Lasix) | | |
| Gabapentin | | |
| Glucophage(Metformin) | | |
| Glucosamine Chondroitin | | |
| Hydrocodone-<br>Acetamenophen | | |
| Ibuprofen (Advil/Motrin) | | |
| Iloprost infusions | | |
| Iron | | |
| Ketorolac tromethamine (Toradol) | | |
| Levemir | | |
| Levothyroxine | | |

| Concomitant Medication | Tofacitinib N=10 n(%) | Placebo N=5<br>n(%) |
|---------------------------|-----------------------|---------------------|
| Lexapro | | |
| Lisinopril(zestril) | | |
| Lopressor | | |
| Loratidine/pseuoephedrine | | |
| Lyrica | | |
| Medical Marijuana | | |
| Methotrexate | | |
| Miralax | | |
| Multi-vitamin | | |
| Mycophenolate-Mofetil | | |
| Neomycin/polyminyx | | |
| Neurontin(Gabapentin) | | |
| Nexium | | |
| Niacin | | |
| Nifedipine(Procardia) | | |
| Normal Saline IV fluids | | |
| Omeprazole(Prilosec) | | |
| Prednisone | | |
| Prevident | | |
| Probiotic | | |
| Ranitidine(Zantac) | | |

| Concomitant Medication | Tofacitinib N=10 n(%) | Placebo N=5<br>n(%) |
|-------------------------|-----------------------|---------------------|
| Riociguat | | |
| Sennosides | | |
| Sildenafil | | |
| Tessalon Perles | | |
| Tesslon Pearls | | |
| Tramadol(Ultram) | | |
| Valacyclovir | | |
| Viagra | | |
| Vicodin | | |
| Vitamin C | | |
| Vitamin D3 | | |
| Vitamin D3 with Calcium | | |
| Voltaren | | |
| Xifaxin | | |
| Zestoretic 20/12.5 | | |
| Zithromax Z-Pak | | |
| alendronate | | |
| amlodipine/olmesartin | | |
| etonogestral Implant | | |
| levothyroxine | | |
| nitrofurantoin | | |

| Concomitant Medication | Tofacitinib N=10<br>n(%) | Placebo N=5<br>n(%) |
|------------------------|--------------------------|---------------------|
| protonix | | |
| riociguat | | |
| trilipix | | |
| zyrtec | | |

[1] The safety population includes all patients randomized to TOFA who received at least one dose of study medication.

Data cutoff date: DDMMYY

# 3.1.2. Safety Analyses

Table 8: TOFA Summary of SAEs by System Organ Class Regardless of Relatedness to Intervention. Safety Population

| Variable | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-------------------------|---------------------|----------------|
| # of SAEs | | |
| # of Subjects with SAEs | | |
| # of Subjects | | |
| SAEs per Subject | | |
| % of Subjects with SAEs | | |

Table 9: TOFA Proportion of Subjects with SAEs by Severity Grade. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Events | | |
| Total Subjects With At Least One Event | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| Grade 4 | | |
| Grade 5 | | |
| Grades 3-5 | | |

# [1] Percentages are 100\*n/N.

The severity grade shown is the greatest grade reported per event for a particular Subject (Grade 1 < Grade 2 < Grade 3 < Grade 4 < Grade 5).

**Listing 3: TOFA Listing of SAEs. Safety Population.** 

| Tro | eatment | Subject<br>ID | SAE# | New SAE<br>since<br>(Date of<br>last<br>report) | SAE Brief<br>Description<br>(Verbatim<br>Term) | Treatment<br>Emergent? | SAE<br>Start<br>Date | SAE<br>Stop<br>Date | Days from<br>Start of<br>Study<br>Medication | Severity<br>Grade | Relationshi<br>p<br>to Study<br>Treatment | Outcome | Study<br>Drug<br>Action<br>Taken | Study Drug<br>Stop Date | Study Drug<br>Start Date |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

There were no SAEs reported as of the data cutoff date.

Treatment emergent adverse events are AEs that are began after the first dose of study medication.

Note: Double-Blind Treatment is expected to last 24 Weeks (168 Days). Those SAEs that started >= Day 169 are assumed to have occurred during the Open Label phase.

Data cutoff date: DDMMYY

**Listing 4: TOFA Listing of Deaths. Safety Population** 

| Treatment | Subject<br>ID | SAE# | New SAE<br>since Aug 4,<br>2017 | SAE<br>Primary<br>Category | SAE<br>Description<br>(Verbatim<br>Term) | Treatment<br>Emergent? | SAE<br>Start<br>Date | SAE<br>Stop<br>Date | Days from<br>Start of<br>Study<br>Medication | Severity<br>Grade | Relationship<br>to Study<br>Treatment | Outcome | Study<br>Drug<br>Action<br>Taken | Treatment<br>Required |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

Conditional Note: There were no deaths reported as of the data cutoff date.

Treatment emergent adverse events are AEs that began after the first dose of study medication.

Table 10: TOFA Proportion of Subjects with Adverse Events by Primary Category. Safety Population.

| Preferred Term | Tofacitinib<br>n (%) [1] | Placebo<br>n (%) [1] |
|---|---|---|
| # of Safety Patients | | |
| # of AEs | | |
| # of Subjects with AEs | | |
| % of Subjects with AEs | | |
| Primary Category | | |
| General Disorders | | |
| Flu-Like Symptoms | | |
| Common Cold | | |
| Weight Gain | | |
| Weight Loss | | |
| Cardiac Disorders | | |
| Tachycardia | | |
| Renal and Urinary Disorders | | |
| Chronic Kidney Disease | | |
| Non-Obstructive Renal Calculi | | |
| Gastrointestinal Disorders | | |
| GERD | | |
| Increased GERD | | |
| Infections and Infestations | | |
| Ulcer Infection | | |

| Preferred Term | Tofacitinib<br>n (%) [1] | Placebo<br>n (%) [1] |
|---|---|---|
| Urinary Tract Infection | | |
| Upper Respiratory Infection | | |
| Otitis Externa | | |
| Investigations | | |
| Hyperkalemia | | |
| Hypercholesterolemia | | |
| Skin and subcutaneous Disorders | | |
| Pruritus (Itching) | | |
| Digital Ulcer Finger | | |
| Nervous System Disorders | | |
| Headache | | |
| Migraine | | |
| Bell's Palsy | | |
| Musculoskeletal and Connective Tissue Disorders | | |
| Joint Pain | | |
| Knee Pain | | |
| Back Pain | | |
| Right Trochanteric Bursitis | | |
| Bilateral Wrist Synovitis | | |
| Respiratory, thoracic and mediastinal disorders | | |
| Maxillary Sinus Inflammation | | |
| Sinus Congestion | | |
| Dyspnea or Exertion | | |

| Preferred Term | Tofacitinib<br>n (%) [1] | Placebo<br>n (%) [1] |
|----------------------|--------------------------|----------------------|
| Vascular Disorders | | |
| Hypertension | | |
| Hypertensive Urgency | | |

[1] Percentages are 100\*n/N. Data cutoff date: DDMMYY

Table 11: TOFA Proportion of Subjects with Adverse Events by Severity. Safety Population.

| Preferred Term | Tofacitinib<br>n (%) [1] | Placebo<br>n (%) [1] |
|------------------------|--------------------------|----------------------|
| # of Safety Patients | | |
| # of AEs | | |
| # of Subjects with AEs | | |
| % of Subjects with AEs | | |
| Severity Grade | | |
| No Adverse Events | | |
| Mild | | |
| Moderate | | |

# [1] Percentages are 100\*n/N.

The severity shown is the greatest reported per event for a particular Subject (Mild < Moderate < Severe).
Data cutoff date: DDMMYY

## Listing 5: TOFA Listing of Treatment Emergent Adverse Events. Safety Population.

| Treatment | Subject<br>ID | New AE<br>Since<br>March<br>5, 2018 | CTCAE Classificaiton | AE Primary<br>Category | AE Start<br>Date | AE End Date | Days from<br>Start of<br>Study<br>Medication | Severity | Relationship<br>to Study<br>Treatment | Outcome | Expected /<br>Unexpected | Study Drug<br>Action<br>Taken | SAE? | Worsening<br>of SSC? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

| Treatment | Subject<br>ID | New AE<br>Since<br>March<br>5, 2018 | CTCAE Classificaiton | AE Primary<br>Category | AE Start<br>Date | AE End Date | Days from<br>Start of<br>Study<br>Medication | Severity | Relationship<br>to Study<br>Treatment | Outcome | Expected /<br>Unexpected | Study Drug<br>Action<br>Taken | SAE? | Worsening<br>of SSC? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

Data cutoff date:DDMMYY

Note: Double-Blind Treatment is expected to last 24 Weeks (168 Days). Those AEs that started >= Day 169 are assumed to have occurred during the Open Label phase.

**Table 12: Adverse Events of Special Interest. Safety Population.** 

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| Total Events | | |
| Total Subjects With At Least One Event | | |
| Herpes Zoster | | |
| Malignancies | | |
| Serious Infections | | |
| Lab Value Abnormalities | | |
| Lymphocytes <500cells mm3 | | |
| ANC <500cells mm3 | | |
| AST/ALT > 3xULN | | |
| Hy's Law Criteria Met | | |
| Hb drop >2gm/dL | | |
| Increase in HDL/LDL > 50% | | |
| Increase in Serum Creatinine > 50% | | |

[1] Percentages are 100\*n/N. Data cutoff date: DDMMYY

The following set of Figures will be of this format:



Figure 1: TOFA Spaghetti Plots of Hemoglobin Over Time by Treatment Figure 2: TOFA Spaghetti Plots of WBC Over Time by Treatment

Figure 3: TOFA Spaghetti Plots of Creatinine Over Time by Treatment

Figure 4: TOFA Spaghetti Plots of Lymphoctyes %Over Time by Treatment

Figure 5: TOFA Spaghetti Plots of Neutrophil % Over Time by Treatment

Figure 6: TOFA Spaghetti Plots of ALT Over Time by Treatment

Figure 7: TOFA Spaghetti Plots of AST Over Time by Treatment

Figure 8: TOFA Spaghetti Plots of Total Cholesterol Over Time by Treatment

Figure 9: TOFA Spaghetti Plots of Triglycerides Over Time by Treatment

Figure 10: TOFA Spaghetti Plots of LDL Over Time by Treatment

Figure 11: TOFA Spaghetti Plots of HDL Over Time by Treatment

Table 13: TOFA Proportion of Subjects with Grade 3 (Severe) or Higher SAEs Within the First 24 Weeks. Primary Outcome. Safety Population.

| Adverse Events | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 3 or Higher Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

[1] Percentages are 100\*n/N.

[2] Poisson Regression, offset for time in study (lesser of 36 weeks or end of study).

Table 14: TOFA Number of Grade 3 (Severe) or Higher SAEs Within the First 24 Weeks. Secondary Outcome. Safety Population.

| Adverse Events | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 3 or Higher SAEs | | |
| Relative Risk [2] | | |
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

[2] Poisson Regression, offset for time in study (lesser of 24 weeks or end of study).

Data cutoff date: 310CT18

Table 15: TOFA Proportion of Subjects with Grade 3 (Severe) or Higher SAEs Within the First 12 Weeks. Secondary Outcome. Safety Population.

| Adverse Events | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 3 or<br>Higher Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

[1] Percentages are 100\*n/N.

[2] Clopper Pearson Exact confidence intervals for proportions with at least a Grade 3 SAE.

[3] Fisher's Exact Test Data cutoff date: DDMMYY

Table 16: TOFA Number of Grade 3 (Severe) or Higher SAEs Within the First 12 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 3 or Higher SAEs | | |
| Relative Risk [2] | | |
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

[1] Percentages are 100\*n/N.

[2] Poisson Regression, offset for time in study (lesser of 12 weeks or end of study).

Table 17: TOFA Proportion of Subjects with Grade 3 (Severe) or Higher SAEs Within the First 36 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 3 or<br>Higher Event | | |

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

[2] Clopper Pearson Exact confidence intervals for proportions with at least a Grade 3 SAE.

[3] Fisher's Exact Test
Data cutoff date: DDMMYY

Table 18: TOFA Number of Grade 3 (Severe) or Higher SAEs Within the First 36 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 3 or Higher SAEs | | |
| Relative Risk [2] | | |
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

[1] Percentages are 100\*n/N.

[2] Poisson Regression, offset for time in study (lesser of 36 weeks or end of study).

Table 19: TOFA Proportion of Subjects with Grade 3 (Severe) or Higher SAEs Within the First 48 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 3 or<br>Higher Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

[2] Clopper Pearson Exact confidence intervals for proportions with at least a Grade 3 SAE.

[3] Fisher's Exact Test

Table 20: TOFA Number of Grade 3 (Severe) or Higher SAEs Within the First 48 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 3 or Higher SAEs | | |
| Relative Risk [2] | | |
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

[2] Poisson Regression, offset for time in study (lesser of 48 weeks or end of study).

Data cutoff date: DDMMYY

Table 21: TOFA Proportion of Subjects with Grade 2 (Moderate) or Higher SAEs Within the First 12 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 2 or<br>Higher Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

[1] Percentages are 100\*n/N.

[2] Clopper Pearson Exact confidence intervals for proportions with at least a Grade 2 SAE.

[3] Fisher's Exact Test

Table 22: TOFA Number of Grade2 (Moderate) or Higher SAEs Within the First 12 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 2 or Higher SAEs | | |
| Relative Risk [2] | | |

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

[2] Poisson Regression, offset for time in study (lesser of 12 weeks or end of study).

Data cutoff date: DDMMYY

Table 23: TOFA Proportion of Subjects with Grade 2 (Moderate) or Higher SAEs Within the First 24 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 2 or<br>Higher Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

[3] Fisher's Exact Test

Table 24: TOFA Number of Grade 2 (Moderate) or Higher SAEs Within the First 24Weeks. Secondary Outcome. Safety Population.

<sup>[2]</sup> Clopper Pearson Exact confidence intervals for proportions with at least a Grade 2 SAE.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 2 or Higher SAEs | | |
| Relative Risk [2] | | |
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

Data cutoff date: DDMMYY

Table 25: TOFA Proportion of Subjects with Grade 2 (Moderate) or Higher SAEs Within the First 36 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 2 or<br>Higher Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

[3] Fisher's Exact Test
Data cutoff date: DDMMYY

<sup>[2]</sup> Poisson Regression, offset for time in study (lesser of 24 weeks or end of study).

<sup>[2]</sup> Clopper Pearson Exact confidence intervals for proportions with at least a Grade 2 SAE.

Table 26: TOFA Number of Grade 2 (Moderate) or Higher SAEs Within the First 36 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 2 or Higher SAEs | | |
| Relative Risk [2] | | |
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

[2] Poisson Regression, offset for time in study (lesser of 36 weeks or end of study).

Table 27: TOFA Proportion of Subjects with Grade 2 (Moderate) or Higher SAEs Within the First 48 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Subjects With At Least One Grade 2 or<br>Higher Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

- [1] Percentages are 100\*n/N.
- [2] Clopper Pearson Exact confidence intervals for proportions with at least a Grade 2 SAE.
- [3] Fisher's Exact Test
  Data cutoff date: DDMMYY

Table 28: TOFA Number of Grade 2 (Moderate) or Higher SAEs Within the First 48 Weeks. Secondary Outcome. Safety Population.

| System Organ Class<br>Preferred Term | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n (%) [1] |
|---|---|---|
| Total Number of Grade 2 or Higher SAEs | | |
| Relative Risk [2] | | |
| 90% Confidence Interval [2] | | |
| p-value [2] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

[2] Poisson Regression, offset for time in study (lesser of 48 weeks or end of study).

Table 29: TOFA Proportion of Subjects with Adverse Events of Special Interest Within the First 12 Weeks.

Secondary Outcome. Safety Population.

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| Total Subjects With At Least One Event | | |
| 90% Confidence Interval [2] | | |

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| p-value [3] | | |
| Herpes Zoster | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Malignancies | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Serious Infections | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Lab Value Abnormalities | | |
| Lymphocytes <500cells mm3 | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| ANC <500cells mm3 | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| AST/ALT > 3xULN | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| Hy's Law Criteria Met | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Hb drop >2gm/dL | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in HDL/LDL > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in Serum Creatinine > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | <u>'</u> |

<sup>[1]</sup> Percentages are 100\*n/N.
[2] Clopper Pearson Exact confidence intervals for proportions with at least of the given AE(s).
[3] Fisher's Exact Test
Data cutoff date: DDMMYY

Table 30: TOFA Proportion of Subjects with Adverse Events of Special Interest Within the First 24 Weeks. Secondary Outcome. Safety Population.

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| Total Subjects With At Least One Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Herpes Zoster | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Malignancies | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Serious Infections | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Lab Value Abnormalities | | |
| Lymphocytes <500cells mm3 | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| ANC <500cells mm3 | | |
| 90% Confidence Interval [2] | | |

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| p-value [3] | | |
| AST/ALT > 3xULN | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Hy's Law Criteria Met | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Hb drop >2gm/dL | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in HDL/LDL > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in Serum Creatinine > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

<sup>[2]</sup> Clopper Pearson Exact confidence intervals for proportions with at least of the given AE(s).
[3] Fisher's Exact Test

Data cutoff date: DDMMYY

Table 31: TOFA Proportion of Subjects with Adverse Events of Special Interest Within the First 36 Weeks. Secondary Outcome. Safety Population.

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| Total Subjects With At Least One Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Herpes Zoster | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Malignancies | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Serious Infections | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Lab Value Abnormalities | | |
| Lymphocytes <500cells mm3 | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| ANC <500cells mm3 | | |
| 90% Confidence Interval [2] | _ | |

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| p-value [3] | | |
| AST/ALT > 3xULN | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Hy's Law Criteria Met | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Hb drop >2gm/dL | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in HDL/LDL > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in Serum Creatinine > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

<sup>[2]</sup> Clopper Pearson Exact confidence intervals for proportions with at least of the given AE(s).
[3] Fisher's Exact Test

Data cutoff date: DDMMYY

Table 32: TOFA Proportion of Subjects with Adverse Events of Special Interest Within the First 48 Weeks. Secondary Outcome. Safety Population.

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| Total Subjects With At Least One Event | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Herpes Zoster | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Malignancies | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Serious Infections | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Lab Value Abnormalities | | |
| Lymphocytes <500cells mm3 | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| ANC <500cells mm3 | | |
| 90% Confidence Interval [2] | | |

| Preferred Term Category | Tofacitinib<br>N=10<br>n (%) [1] | Placebo<br>N=5<br>n(%) [1] |
|---|---|---|
| p-value [3] | | |
| AST/ALT > 3xULN | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Hy's Law Criteria Met | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Hb drop >2gm/dL | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in HDL/LDL > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |
| Increase in Serum Creatinine > 50% | | |
| 90% Confidence Interval [2] | | |
| p-value [3] | | |

<sup>[1]</sup> Percentages are 100\*n/N.

<sup>[2]</sup> Clopper Pearson Exact confidence intervals for proportions with at least of the given AE(s).
[3] Fisher's Exact Test

Data cutoff date: DDMMYY

Table 33: TOFA Labs Over Time. Safety Population [1]

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------------|-----------|----------|---------------------|----------------|
| Hemoglobin | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------------|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Hematocrit | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----------|-----------|----------|---------------------|----------------|
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Platelets | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| RBC | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| WBC | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-------------|-----------|----------|---------------------|----------------|
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Neutrophils | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | _ |
| | Baseline | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-------------|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Lymphocytes | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----------|-----------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Monocytes | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|----------|----------|---------------------|----------------|
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-------------|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Eosinophils | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----------|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Basophils | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|----------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|--------|-----------|----------|---------------------|----------------|
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Sodium | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|----------|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Chloride | Screening | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----------|-----------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Potassium | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| AST | Screening | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| ALT | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | Min, Max | | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|-----------|----------|---------------------|----------------|
| Glucose | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | Mean(SD) | | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Calcium | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------------|-----------|----------|---------------------|----------------|
| | | Min, Max | | |
| Creatinine | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------|-----------|----------|---------------------|----------------|
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| eGFR | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| | | Median | | |
| | | Min, Max | | |
| Total Bilirubin | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| BUN | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------------|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Total Protein | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Albumin | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Alkaline<br>Phosphatase | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | _ | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| ESR | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| CRP | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Total Cholesterol | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| HDL | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| LDL | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------------|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| Triglycerides | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

[1] The safety population includes all patients randomized to TOFA who received at least one dose of study medication.

Note: Lipid panel only done at Screening and Weeks 6, 30, and 36. Data cutoff date: DDMMYY

**Table 34: TOFA Vital Signs Over Time. Safety Population [1]** 

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|----------------|-----------|----------|---------------------|----------------|
| Temperature(C) | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Respiratory Rate | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Systolic Blood<br>Pressure | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Diastolic Blood<br>Pressure | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | _ |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|----------|----------|---------------------|----------------|
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-------|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Pulse | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------------|-----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Height(cm) | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|----------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------------|-----------|----------|---------------------|----------------|
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| Weight(kg) | Screening | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|-----------|----------|---------------------|----------------|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| BMI | Screening | N | | |
| | | Mean(SD) | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|----------|----------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | Baseline | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 6 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 30 | N | | |
| | | Mean(SD) | | |
| | | Median | | |

| Lab | Time | Status | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|----------|---------------------|----------------|
| | | Min, Max | | |
| | Week 36 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |

Data cutoff date: DDMMYY

<sup>[1]</sup> The safety population includes all patients randomized to TOFA who received at least one dose of study medication.

Table 35: TOFA Physical Examination Findings. Safety Population [1]

| Body System | Time | Tofacitini<br>b<br>N (%) | Placebo<br>N (%) |
|---|---|---|---|
| Head Eyes Ears Nose and<br>Throat | Screening | | |
| | Week 6 | | |
| | Week 12 | | |
| | Week 24 | | |
| Respiratory | Screening | | |
| | Week 6 | | |
| | Week 12 | | |
| Cardiovascular | Screening | | |
| | Week 12 | | |
| | Week 24 | | |
| | Week 30 | | |
| Abdomen | Screening | | |
| | Week 6 | | |
| | Week 24 | | |
| Musculoskeletal | Screening | | |
| | Week 6 | | |
| | Week 12 | | |

| Body System | Time | Tofacitini<br>b<br>N (%) | Placebo<br>N (%) |
|----------------|-----------|--------------------------|------------------|
| | Week 24 | | |
| | Week 30 | | |
| Dermatological | Screening | | |
| | Week 6 | | |
| | Week 12 | | |
| | Week 24 | | |
| | Week 30 | | |
| | Week 36 | | |
| | Week 48 | | |

Note: Percentages are based on the number of subjects with abnormal findings in the Safety Population. [1] The Safety Population includes all randomized subjects who received at least one dose of study medication. Data cutoff date: DDMMYY

## 3.1.3. Efficacy Analyses

**Table 36: TOFA Change From Baseline in mRSS Total Score. ITT Population** 

| Status | Tofacitinib<br>N=10 | Placebo<br>N= 5 |
|---------|---------------------|-----------------|
| Week 12 | | |
| N | | |

| Status | Tofacitinib<br>N=10 | Placebo<br>N= 5 |
|-------------|---------------------|-----------------|
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value [2] | | |
| Week 24 | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value [2] | | |
| Week 36 | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value [2] | | |
| Week 48 | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |

| Status | Tofacitinib<br>N=10 | Placebo<br>N= 5 |
|-------------|---------------------|-----------------|
| p-value [2] | | |

- [1] The ITT population includes all patients randomized to TOFA.[2] Two-sample t-tests

Data cutoff date: DDMMYY

**Table 37: TOFA Responder Status Relative to Baseline in mRSS Total** Score. ITT Population [1]

| Status | Tofacitinib<br>N=10<br>n(%) | Placebo<br>N= 5<br>n(%) | p-value<br>[2] |
|---|---|---|---|
| Week 12 | | | |
| At least 20% Reduction | | | |
| At least 40% Reduction | | | |
| At least 60% Reduction | | | |
| Week 24 | | | |
| At least 20% Reduction | | | |
| At least 40% Reduction | | | |
| At least 60% Reduction | | | |

[1] The ITT population includes all patients randomized to TOFA. [2] Fisher's Exact Test

Data cutoff date: DDMMYY

Table 38: TOFA Change From Baseline in mRSS Scores. ITT Population [1]

| Variable [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|----------------------|---------------------|----------------|
| Week 12 | | |
| Total Score | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value [2] | | |
| Representative Score | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value [2] | | |
| Maximum Score | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value | | |

| Variable [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|----------------------|---------------------|----------------|
| Week 24 | | |
| Total Score | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value | | |
| Representative Score | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value | | |
| Maximum Score | | |
| N | | |
| Mean(SD) | | |
| Median | | |
| Min, Max | | |
| p-value | | |

**Table 39: TOFA Change From Baseline in Physician Global Health Assessment. ITT Population [1]** 

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| Week 12 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 36 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 48 | N | | |

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------|---------------|---------------------|----------------|
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |

**Table 40: TOFA Change From Baseline in Patient Global Health Assessment. ITT Population [1]** 

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| Week 12 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| | p-value | | |
| Week 36 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 48 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |

[1] The ITT population includes all patients randomized to TOFA.[2] Two-sample t-testsData cutoff date: DDMMYY

Table 41: TOFA Change From Baseline in Health-Related Quality of Life (HRQOL) using PROMIS-29. ITT Population [1]

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| Week 12 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 36 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 48 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------|---------------|---------------------|----------------|
| | p-value | | |

[2] Two-sample t-tests
Data cutoff date: DDMMYY

Table 42: TOFA Change From Baseline in Scleroderma Health assessment Questionnaire-Disability Index (SHAQ-DI). ITT Population [1]

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| Week 12 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 36 | N | | |

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 48 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |

Table 43: TOFA Change From Baseline in UCLA SCTC Gastrointestinal Symptoms Total Score. ITT Population [1]

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| Week 12 | N | | |
| | Mean(SD) | | |
| | Median | | |

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| | Min, Max | | |
| | p-value | | |
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 36 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 48 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | _ | |
| | p-value | | |

<sup>[1]</sup> The ITT population includes all patients randomized to TOFA.[2] Two-sample t-testsData cutoff date: DDMMYY

Table 44: TOFA Change From Baseline in Scleroderma-Related Skin Symptoms Assessed by PRO-SRSS. ITT Population [1]

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|---------------|---------------------|----------------|
| Week 12 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 36 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value | | |
| Week 48 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |

| Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------|---------------|---------------------|----------------|
| | p-value | | |

Table 45: TOFA Change From Screening in PFTs. ITT Population [1]

| PFT | Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| % Predicted FVC | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| | Week 48 | N | | |

| PFT | Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---|---|---|---|---|
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| % Predicted FEV | Week 12 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| % Predicted DLCO | Week 12 | N | | |
| | | Mean(SD) | | |

| PFT | Time | Statistic [2] | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|-----|---------|---------------|---------------------|----------------|
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| | Week 24 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |
| | Week 48 | N | | |
| | | Mean(SD) | | |
| | | Median | | |
| | | Min, Max | | |
| | | p-value | | |

[1] The ITT population includes all patients randomized to TOFA.[2] Two-sample t-testsData cutoff date: DDMMYY

Table 46: TOFA Change From Screening to Week 24 in Left Ejection Fraction (Maximum of Range). ITT Population [1]

| Time | Statistic | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|-------------|---------------------|----------------|
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |
| | p-value [2] | | |

Table 47: TOFA Change From Screening to Week 24 in Tricuspid Regurgitation Jet. ITT Population [1]

| Time | Statistic | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|---------|-----------|---------------------|----------------|
| Week 24 | N | | |
| | Mean(SD) | | |
| | Median | | |
| | Min, Max | | |

| Time | Statistic | Tofacitinib<br>N=10 | Placebo<br>N=5 |
|------|----------------|---------------------|----------------|
| | p-value<br>[2] | | |

[1] The ITT population includes all patients randomized to TOFA.[2] Two-sample t-testsData cutoff date: DDMMYY